CLINICAL TRIAL: NCT03262285
Title: Corneal Endothelial Cell Loss After Phacoemulsification Compared With Extracapsular Cataract Extraction in Management of Senile Cataract
Brief Title: Corneal Endothelial Cell Loss After Phacoemulsification Compared With Extracapsular Cataract Extraction
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rawda Abdelnaser, resident, Assiut University
Other Study IDs: CECLPEECCE
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-05

CONDITIONS: Senile Cataract
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- phacoemulsification: patients undergoing phacoemulsification surgery for senile cataract
  Interventions: Procedure: phacoemulsification
- extracapsular cataract extraction: patients undergoing extracapsular cataract extraction surgery for senile cataract
  Interventions: Procedure: extracapsular cataract extraction

INTERVENTIONS:
Procedure: phacoemulsification — removal of cataract using ultrasound waves
  Groups: phacoemulsification
Procedure: extracapsular cataract extraction — removal of cataract using surgical corneal incision
  Groups: extracapsular cataract extraction

SUMMARY:
the investigators will compare between the endothelial cell loss after phacoemulsification and extracapsular cataract extraction in management of senile cataract

DETAILED DESCRIPTION:
Age related cataract is believed to be the main cause of reversible blindness worldwide and in developing countries. Population-based studies have reported that cataract is responsible for 47.8% to 51% of all global blindness.

Several studies compared phacoemulsification and conventional extracapsular cataract extraction regarding several aspects such as postoperative inflammation and visual rehabilitation. studies proved that phacoemulsification has faster rehabilitation ,less astigmatism and better postoperative vision .However, Extracapsular cataract extraction is still the operation of choice in some cataract cases.

The normal corneal endothelium is a single layer of uniformly sized cells with a predominantly hexagonal shape. Adult density of approximately 2400 - 3200 cells/mm².The number of cells decreases at about 0.6% per year and neighbouring cells enlarge to fill the space as the cells cannot regenerate.The minimum cell density necessary for adequate function is in the range of 400 to 700 cells/mm2.

The effect of cataract surgery on corneal endothelium is an important factor that affects postoperative vision .However, it is accepted all over the world that there is definite loss of some endothelial cells with all techniques of cataract surgery. Previously, cataract surgery caused enormous loss of endothelial cells , but with enhancement of equipment and surgical techniques, cataract surgery today results in 6-14%loss of endothelial cells.

Specular microscopy is a noninvasive photographic technique that allows visualization and analysis of corneal endothelium. specular microscopy is used to show cell count and cell shape in the scanned area.

ELIGIBILITY:
Inclusion Criteria:

* Cases of senile cataract of both sexes will be included in this study

Exclusion Criteria:

* Corneal endothelial pathologies such as Fuch's dystrophy
* Complicated cataract
* Cataract with history of trauma
* Coexisting eye pathology

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with senile cataract
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
percentage of endothelial cell loss | 5 minutes
  specular microscopy will be done to measure the endothelial cell count before and after the intervention to measure the percentage of loss

SECONDARY OUTCOMES:
changes in shape of endothelial cell | 5 minutes
  specular microscopy will be done to identify changes in hexagonality of endothelial cells after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ryad, professor, Study Chair — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Lundstrom M, Goh PP, Henry Y, Salowi MA, Barry P, Manning S, Rosen P, Stenevi U. The changing pattern of cataract surgery indications: a 5-year study of 2 cataract surgery databases. Ophthalmology. 2015 Jan;122(1):31-8. doi: 10.1016/j.ophtha.2014.07.047. Epub 2014 Sep 16. PMID 25234011
- [Background] Bourne RR, Stevens GA, White RA, Smith JL, Flaxman SR, Price H, Jonas JB, Keeffe J, Leasher J, Naidoo K, Pesudovs K, Resnikoff S, Taylor HR; Vision Loss Expert Group. Causes of vision loss worldwide, 1990-2010: a systematic analysis. Lancet Glob Health. 2013 Dec;1(6):e339-49. doi: 10.1016/S2214-109X(13)70113-X. Epub 2013 Nov 11. PMID 25104599
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Wang W, Yan W, Muller A, He M. A Global View on Output and Outcomes of Cataract Surgery With National Indices of Socioeconomic Development. Invest Ophthalmol Vis Sci. 2017 Jul 1;58(9):3669-3676. doi: 10.1167/iovs.17-21489. PMID 28728174
- [Background] Gogate PM, Kulkarni SR, Krishnaiah S, Deshpande RD, Joshi SA, Palimkar A, Deshpande MD. Safety and efficacy of phacoemulsification compared with manual small-incision cataract surgery by a randomized controlled clinical trial: six-week results. Ophthalmology. 2005 May;112(5):869-74. doi: 10.1016/j.ophtha.2004.11.055. PMID 15878068
- [Background] Bourne WM, Nelson LR, Hodge DO. Central corneal endothelial cell changes over a ten-year period. Invest Ophthalmol Vis Sci. 1997 Mar;38(3):779-82. PMID 9071233
- [Background] Bourne RR, Minassian DC, Dart JK, Rosen P, Kaushal S, Wingate N. Effect of cataract surgery on the corneal endothelium: modern phacoemulsification compared with extracapsular cataract surgery. Ophthalmology. 2004 Apr;111(4):679-85. doi: 10.1016/j.ophtha.2003.07.015. PMID 15051198
- [Background] Trnavec B, Cuvala J, Cernak A, Vodrazkova E. [Comparison of corneal endothelial cells after ECCE and phacoemulsification of the lens]. Cesk Slov Oftalmol. 1997 Aug;53(4):240-3. Slovak. PMID 9377317